CLINICAL TRIAL: NCT05171543
Title: Effect of Combined Use of an Allograft and a Membrane on the Healing Outcome of Apicomarginal Defects Using 2D and 3D Evaluation
Brief Title: Effect of Combined Use of an Allograft and Membrane on the Healing Outcome of Apicomarginal Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Rahul Sharma
Record Dates: First submitted 2021-12-10; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-05

CONDITIONS: Apicomarginal Defects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periapical surgery with placement of an allograft and a membrane (Experimental): Patients will undergo periapical surgery and an allograft and a membrane will be placed inside the bony crypt and over the denuded root surface respectively before closure of the flap.
  Interventions: Procedure: Periapical surgery with placement of an allograft and a membrane
- Periapical surgery with no placement of any graft or membrane (No Intervention): Patients will undergo periapical surgery with no placement of any graft or membrane in the control group.

INTERVENTIONS:
Procedure: Periapical surgery with placement of an allograft and a membrane — Periapical surgery will be done followed by placement of an allograft into the defect and a membrane over the defect before closure of the flap.
  Arms: Periapical surgery with placement of an allograft and a membrane

SUMMARY:
Healing of apicomarginal defects using 2 different groups, one being treated with the use of an allograft and a membrane and a control group, will be assessed and compared using 2D and 3D criteria. Also,quality of life will be compared between the two groups.

DETAILED DESCRIPTION:
Periapical surgery is a viable treatment option in teeth with persistent apical periodontitis, especially in cases which fail to heal by non surgical treatment. Kim and Kratchman classified periradicular lesions into categories A-F. Lesions A-C are of endodontic origin without any periodontal pockets and vary with respect to the size of periapical radiolucency while D-F are combined endodontic - periodontal origin and are ranked accoding to the magnitude of periodontal breakdown. Type F defects are commonly referred to as apicomarginal defects and have worst prognosis among all. The lower success rate is attributed to the apical migration of junctional epithelium and intrusion of non osteogenic connective tissue into the periapical region.

Various resorbable and non resorbable collagen membrane with or without xenograft, allograft and alloplastic materials have been used in different studies. Although animal studies have reported high success rates with the use of bone graft materials and membranes over the controls but no human study till date has evaluated or compared the effect of using an allograft and membrane versus Control.

Thus, the aim of the present study is to investigate to two hypothesis. The first null hypothesis stated that there would be no difference between quality of life and healing outcome of periapical defects with periodontal communications following surgery using membrane with allograft and the conventional control group utilizing no GTR technique. The second null hypothesis stated that there would be no difference in outcome derived from the assessment of 2D periapical radiographs and 3D CBCT imaging.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 16 years and older consenting to the surgical procedure as well as agreeing to preoperative and at least 1 follow-up CBCT evaluation after 12 months 2. Noncontributory medical history (American Society of Anesthesiologists class I and II) 3. Patients with a deep narrow pocket with probing depth >6 mm confined to buccal aspect of the root, 4. Negative response to vitality tests, 5. Radiographic evidence of radiolucency, 6. Failed previous root canal treatment and retreatment at least 1 year previously, 7. Previous surgery with unresolved bony lesion, 8. Recurrent episodes of purulent discharge, and 9. Adequate final restoration with no clinical evidence of coronal leakage.

Exclusion Criteria:

- 1. Patients with medical history with American Society of Anesthesiologists class III to V or Any systemic disease contraindicating oral surgical procedures, potentially affecting the healing process.

2. Chronic generalized periodontitis, 3. Evidence of root fracture, 4. resorptive processes involving more than apical third of the root

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Healing of apicomarginal defects. | Baseline to 12 months
  Patients will be checked clinically for absence of signs and symptoms. Radiographic 2D assessment will be done by Rud and Molven criteria as follows:-
  Complete healing- defined by re-establishment of the lamina dura Incomplete healing (scar tissue) Uncertain healing Unsatisfactory healing (failure). 3D healing will be assessed by modified PENN 3D criteria(Schloss et al) as-
  Complete healing Limited healing Uncertain healing Unsatisfactory healing.

SECONDARY OUTCOMES:
Assessment of quality of life | Baseline to day 7 postoperatively
  All patients will be given a questionnaire (Igor Tsesis et al) with 15 questions to evaluate their quality of life for 7 days postsurgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanjay Tewari, Rohtak, Haryana, India